CLINICAL TRIAL: NCT06317233
Title: Outcomes of a Longitudinal Multidisciplinary Program for the Treatment of Chronic Pelvic Pain, Incorporating Online and Mobile Applications to Promote Self Efficacy
Brief Title: Outcomes of a Multidisciplinary Program for the Treatment of Chronic Pelvic Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007131
Record Dates: First submitted 2024-03-04; First posted 2024-03-19 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pelvic Pain Syndrome
Keywords: treatment guide; patient satisfaction; pain scores
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention)
- Treatment Guide plus Standard of Care (Experimental)
  Interventions: Behavioral: Chronic Pelvic Pain Treatment Guide

INTERVENTIONS:
Behavioral: Chronic Pelvic Pain Treatment Guide — The treatment guide includes mobile and web-based resources and applications specifically chosen to empower patients with information and to promote self-efficacy. The treatment guide is designed to be easily understood, visually appealing, and largely translatable from institution to institution. Patients using the treatment guide will be followed with a clearly defined follow up schedule, which includes touch points between appointments to aid with resource navigation.
  Arms: Treatment Guide plus Standard of Care

SUMMARY:
The goal of this clinical trial is to test the impact of a detailed treatment handbook and follow-up schedule on women seeking care for chronic pelvic pain in a gynecology office-based practice. The main questions it aims to answer are:

* How does the handbook and follow-up impact patient satisfaction?
* How does the handbook and follow-up impact patient pain and quality of life scores? Participants will be randomized to receive the office standard of care, or standard of care plus a printed handbook customized to highlight their diagnosis, treatment plan and follow-up schedule.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is a common and multi-factorial condition resulting in high physical, emotional and psychological burden for patients. Multimodal treatments have been shown to be most effective in addressing the multifactorial nature of CPP, but remain challenging for patients and providers to navigate. Investigators have created a CPP treatment guide which clearly defines resources and management strategies in an effort to help patients understand their own diagnosis, treatment options and follow up schedule. The treatment guide includes mobile and web-based resources and applications specifically chosen to empower patients with information and to promote self-efficacy. The treatment guide is designed to be easily understood, visually appealing, and largely translatable from institution to institution. Patients using the treatment guide will be followed with a clearly defined follow up schedule, which includes touch points between appointments to aid with resource navigation. The investigators hypothesize that patients with CPP who are provided our treatment guide will experience improved satisfaction with their care, in addition to improved quality of life measures and pain scores as compared to those who undergo standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 or older
* Diagnosis of chronic pelvic pain

Exclusion Criteria:

* Primary language other than English
* Pregnancy
* Inability to attend follow-up appointment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-06 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | at several intervals over the course of 1 year
  Measured using the Patient Satisfaction Questionnaire Short Form (PSQ-18). The PSQ-18 yields separate scores for each of seven different subscales: general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, accessibility and convenience. The items are scored so that high scores reflect satisfaction with medical care on a 1-5 scale.

SECONDARY OUTCOMES:
Pain Catastrophizing | at several intervals over the course of 1 year
  Measured using the Pain Catastrophizing Scale which includes 13 questions scored from 0-4, with a minimum score of 0 and maximum score of 52. A higher score reflects a greater degree of pain catastrophizing.
Pelvic Pain | at several intervals over the course of 1 year
  Measured using a validated pelvic pain specific questions, with responses ranging from 0-10, for a minimum score of 0 and maximum score of 50. A higher score reflects a greater degree of pelvic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT06317233/Prot_000.pdf